CLINICAL TRIAL: NCT02338583
Title: A Prospective, Multi-Center Evaluation of a Powered Surgical Stapler in Video-Assisted Thoracoscopic Lung Resection Procedures in China
Brief Title: Powered Surgical Stapler in VATS Lung Resection Procedures in China
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC-14-003
Record Dates: First submitted 2015-01-12; First posted 2015-01-14 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Echelon Flex™ 45 and 60 Powered ENDOPATH® Stapler Articulating Endoscopic Linear Cutter

SUMMARY:
This prospective, single-arm multi-center study will provide clinical data in an observational setting using the Echelon Flex™ 45 and 60 Powered ENDOPATH® Stapler Articulating Endoscopic Linear Cutters (study Endocutter). Individuals undergoing VATS lobectomy for suspected or confirmed Non Small Cell Lung Cancer (NSCLC), or individuals undergoing VATS diagnostic wedge resection in accordance with their institution's Standard of care (SOC), and who meet study entry criteria, may be enrolled.

Study procedures will include a wedge resection, wedge resection followed by lobectomy of the same lobe, or lobectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed of NSCLC (up to and including Stage II), or individuals undergoing VATS diagnostic wedge resection in accordance with their institution's Standard of care (SOC);
2. Scheduled for lung resection surgery (lobectomy or wedge resection) involving only one lobe of the lung;
3. Performance status 0-1 (Eastern Cooperative Oncology Group classification);
4. ASA score < 3;
5. No prior history of VATS or open lung surgery;
6. Willing to give consent and comply with study-related evaluation and treatment schedule; and
7. At least 18 years of age.

Exclusion Criteria:

Subjects satisfying the following criteria will be eligible for participation in this study:

1. Suspected or confirmed of NSCLC (up to and including Stage II), or individuals undergoing VATS diagnostic wedge resection in accordance with their institution's Standard of care (SOC);
2. Scheduled for lung resection surgery (lobectomy or wedge resection) involving only one lobe of the lung;
3. Performance status 0-1 (Eastern Cooperative Oncology Group classification);
4. ASA score < 3;
5. No prior history of VATS or open lung surgery;
6. Willing to give consent and comply with study-related evaluation and treatment schedule; and
7. At least 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals scheduled for VATS lobectomy or diagnostic VATS wedge resection in accordance with their institution's SOC
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of prolonged air leaks | 30 days

SECONDARY OUTCOMES:
2.Occurrence of postoperative air leaks | 30 days
Length of stay (LOS) | 30 days
Volume of estimated intra-operative blood loss | Intra-operative
5.Time to chest tube removal | 30 days

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing
  - Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing
  - Wuhan Tongji Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
via publication